CLINICAL TRIAL: NCT00046748
Title: Ph III, 28-wk, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess Efficacy, Safety, Tolerability of SC Omalizumab in Adults and Adolescents w/ Severe Persist. Allergic Asthma & Are Inadequately Controlled Despite GINA (2002) Step 4 Tx
Brief Title: Efficacy and Safety of Omalizumab in Patients With Severe Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025A2306
Record Dates: First submitted 2002-10-02; First posted 2002-10-04 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

INTERVENTIONS:
Drug: Omalizumab

SUMMARY:
The purpose of this study is to determine the effect of omalizumab, compared to placebo, on clinically significant asthma exacerbation rates in adolescents and adults with asthma.

ELIGIBILITY:
* with the diagnosis of allergic asthma >1 year duration who, in addition to the standards of the American Thoracic Society (ATS) meet the following criteria:
* with a positive prick skin test (diameter of wheal > 3 mm) to at least one perennial allergen (e.g. dust mite, animal dander, cockroaches), within the past 5 years or at Visit 1, to which the patient will be exposed on a regular basis (most days) for the duration of the study. A RAST test may be performed for patients with a borderline skin prick test result.
* with total serum IgE level 30 to 700 IU/ml.
* demonstrating 12% increase in FEV1 over baseline value within 30 minutes of taking up to 4 puffs salbutamol (albuterol) or nebulized salbutamol up to 5mg (or equivalent of alternative B-2 agonist) documented within the past year, at screening, during the run-in period or at baseline prior to randomization.
* with FEV1 40-80% of predicted normal value for the patient (demonstrable at least 6 hours after short acting B-2 agonist use or 12 hours after long acting B-2 agonist use) at baseline.
* who have either experienced at least two independent asthma exacerbations requiring unscheduled clinical intervention with a systemic corticosteroid in the past year.

or:

* been admitted to hospital (including intensive care unit) or received emergency room (including urgent care centers) treatment in the past 12 months for an asthma exacerbation, which in accordance with the GINA guidelines met all of the following criteria for a severe exacerbation:

  1. PEF or FEV1< 60% of predicted/personal best, or patient is too breathless to provide PEF.
  2. No improvement after initial treatment and therefore requiring repeated treatment with inhaled B-2 agonist (high dose, spacer or nebulized).
  3. Requiring treatment with systemic corticosteroids
* receiving high dose inhaled corticosteroid (at least 1000ug beclomethasone dipropionate or equivalent) and a regular inhaled long acting B-2 agonist for at least 3 months prior to screening and prior to at least two independent asthma exacerbations requiring unscheduled clinical intervention with a systemic corticosteroid in the past year or the severe asthma exacerbation requiring the hospitalization/ER visit.
* who are receiving an ICS dosage > 1000ug beclomethasone dipropionate or equivalent and a regular inhaled long acting B-2 agonist for the last 4 weeks of the run-in period and at randomization (to be maintained throughout the study).
* whose asthma medication remains unchanged in the final 4 weeks of the run-in period (to be maintained throughout the study).
* with evidence of poor asthma symptom control at screening (based on patient history) and during the 4 weeks immediately prior to baseline.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2001-12; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Clinically significant asthma exacerbation

SECONDARY OUTCOMES:
Medical resource utilization
Time to first asthma exacerbation
Quality of Life assessment at baseline, last visit
Frequency of asthma rescue medication use
Safety/tolerability of omalizumab

REFERENCES:
- [Derived] Chen M, Choo E, Yoo B, Raut P, Haselkorn T, Pazwash H, Holweg CTJ, Hudes G. No difference in omalizumab efficacy in patients with asthma by number of asthma-related and allergic comorbidities. Ann Allergy Asthma Immunol. 2021 Jun;126(6):666-673. doi: 10.1016/j.anai.2021.01.015. Epub 2021 Jan 17. PMID 33465457
- [Derived] Busse WW, Szefler SJ, Haselkorn T, Iqbal A, Ortiz B, Lanier BQ, Chipps BE. Possible Protective Effect of Omalizumab on Lung Function Decline in Patients Experiencing Asthma Exacerbations. J Allergy Clin Immunol Pract. 2021 Mar;9(3):1201-1211. doi: 10.1016/j.jaip.2020.10.027. Epub 2020 Oct 24. PMID 33223095
- [Derived] Busse WW, Humbert M, Haselkorn T, Ortiz B, Trzaskoma BL, Stephenson P, Garcia Conde L, Kianifard F, Holgate ST. Effect of omalizumab on lung function and eosinophil levels in adolescents with moderate-to-severe allergic asthma. Ann Allergy Asthma Immunol. 2020 Feb;124(2):190-196. doi: 10.1016/j.anai.2019.11.016. Epub 2019 Nov 22. PMID 31760132